CLINICAL TRIAL: NCT05556941
Title: Development and Efficacy of Metacognitive Intervention for Individuals With Severe Mental Disorders
Brief Title: Metacognitive Intervention for Individuals With Severe Mental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Naomi Josman, Prof, University of Haifa
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Kaizerman-Dinerman2022
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Schizophrenia
Keywords: Executive function; Meta-cognition; Schizophrenia; Meta-cognitive intervention
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Before and after intervention
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metacognitive Group Intervention (Experimental): Meta cognitive intervention protocol based on the dynamic interactional model of cognition (Toglia, 2005), and specifically tailored to individuals with schizophrenia.
  Interventions: Behavioral: Metacognitive Group Intervention
- Occupational therapy standard care (Active Comparator): Standard care of occupational therapy in mental health, focused on work occupations.
  Interventions: Behavioral: Occupational therapy standard care

INTERVENTIONS:
Behavioral: Metacognitive Group Intervention — The investigators developed an initial Meta cognitive group intervention protocol based on the dynamic interactional model of cognition (Toglia, 2005), and specifically tailored it to individuals with schizophrenia.
  Arms: Metacognitive Group Intervention
Behavioral: Occupational therapy standard care — Occupational therapy standard care
  Arms: Occupational therapy standard care

SUMMARY:
The overall aim of this study was to develop a meta-cognitive group intervention in order to apply it and to understand and distinguish the components that influence participation among people with schizophrenia

DETAILED DESCRIPTION:
The overall aim of this study was to develop a Meta cognitive group intervention in order to apply it and to understand and distinguish the components that influence participation among people with schizophrenia. The specific objectives were to:

1. Improve participation by increasing the effectiveness of cognitive strategy use and teaching clients to independently review performance and to examine the strategy's effectiveness.
2. Compare the use of cognitive strategies between participants with schizophrenia and their matched controls following the Meta cognitive group intervention and to correlate the cognitive strategies use and participation following the Meta cognitive group.
3. Examine whether symptoms moderate the association between metacognitive outcomes and participation among people with schizophrenia following the Meta cognitive group.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of schizophrenia by a licensed psychiatrist
* Fluency in Hebrew
* t-score of at least 65 on the Behavior Rating Inventory of Executive Function-Adult version

Exclusion Criteria:

* Severe psychiatric hospitalization of over 24 hours during the month prior to the beginning of the study
* Used drugs or alcohol

Ages: 23 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | 15 minutes
  The Positive and Negative Syndrome Scale is a 30-item scale with seven positive and seven negative symptoms items and 16 psychopathological items. The severity of each item is rated on a scale from 1 (none) to 7 (most severe). A general Positive and Negative Syndrome Scale score is between 30 (lack of symptoms) and 210 (very severe state of the disease). Potential ranges are 7 to 49 for the positive and negative symptom scales and from 16 to 12 for the general psychopathology scale.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Josman, PhD, Principal Investigator — University of Haifa

IPD SHARING:
Plan to Share IPD: No
In accordance with the Helsinki Declaration and University ethical committee principles, the data used in this study cannot be made available because it was not anonymous.

REFERENCES:
- [Result] Kaizerman-Dinerman A, Roe D, Josman N. An efficacy study of a metacognitive group intervention for people with schizophrenia. Psychiatry Res. 2018 Dec;270:1150-1156. doi: 10.1016/j.psychres.2018.10.037. Epub 2018 Oct 13. PMID 30482631
- [Result] Kaizerman-Dinerman A, Josman, Roe D. The use of cognitive strategies among people with schizophrenia: a randomized comparative study. The Open Journal of Occupational Therapy. 2019; 7(3): 1-12.
- [Derived] Kaizerman-Dinerman A, Roe D, Demeter N, Josman N. Do symptoms moderate the association between participation and executive functions outcomes among people with schizophrenia? BMC Psychiatry. 2023 Jan 17;23(1):42. doi: 10.1186/s12888-022-04510-0. PMID 36650458